CLINICAL TRIAL: NCT03036345
Title: Prediction of Post-operative Cognitive Decline Following Shoulder Surgery in the Beach Chair Position: The Value of Cerebral Oximetry
Brief Title: Cerebral Perfusion in the Beach Chair Position
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Brisbane Hand and Upper Limb Research Institute (Other)
Collaborators: Medtronic (Industry); CAS Medical Systems, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ISR-2016-10757
Record Dates: First submitted 2016-12-29; First posted 2017-01-30 (Estimated); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Cognitive Dysfunction
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Surgery patients (Experimental): Patients receiving shoulder surgery in the Beach Chair Position, and monitored by both INVOS and FORE-SIGHT monitors.
  Interventions: Device: Dual-monitoring

INTERVENTIONS:
Device: Dual-monitoring — Monitored using both INVOS and FORE-SIGHT monitors.

SUMMARY:
Surgery to the shoulder may be performed with patients seated upright in a position known as the "Beach Chair Position (BCP)." This position has certain advantages compared to alternative surgical positions (e.g. side lying) in some situations. However, it has been found that surgery in the BCP can temporarily decrease the amount of oxygen in the brain as a result of the combined effects of gravity and anaesthesia. This can result in complications following surgery such as some memory loss and confusion. Rarely, more serious complications have been reported in the past including death and stroke.

Due to these reported complications the use of "cerebral oximetry" during shoulder surgery in the BCP has become more common. Before and during surgery, a monitor placed on the patients forehead measures the amount of oxygen present in the brain to help control this to an acceptable level. A number of monitors are now commercially available. Two monitors are commonly discussed in the literature; the INVOS™ 5100 and the FORE-SIGHT® machines. However, the actual relationship between the supply of oxygen to the brain during surgery and the chance of later developing problems with memory and thinking (known as "post operative cognitive decline" - POCD) is not clear. It is also not known if one monitor is more accurate than another at predicting these complications.

Therefore, the main aim of this study is to examine the relationship between cerebral oxygen levels during shoulder surgery and the incidence of POCD (i.e. problems with memory and thinking). A second aim is to compare the INVOS™ 5100 and FORE-SIGHT® monitors ability to measure cerebral oxygen and cerebral desaturation events (CDEs) as well as the importance of other key clinical variables (e.g. blood pressure, nausea, body fat etc).

DETAILED DESCRIPTION:
PURPOSE OF THE INVESTIGATION The purpose of this investigation is to generate evidence about cerebral oxygenation during shoulder surgery and the incidence of POCD. Currently, evidence relating to POCD following surgery is conflicting and relates mostly to outcomes following cardiac surgery. There is a strong need to explore this relationship in the specific context of shoulder surgery in the BCP.

INTERVENTION GROUPS This study will involve a single prospective cohort. Patients who meet the selection criteria will be recruited to the study following voluntary informed consent . Cerebral oxygenation will be measured by application of cerebral oximeters to each patients forehead.

AIM OF THE STUDY This study has three aims; (i) To examine the relationship between cerebral desaturation during shoulder surgery in the BCP, and the incidence of POCD.

(ii) To determine the variation in cerebral oxygenation recorded using randomised (for superior/inferior) simultaneous application of the INVOS™ and FORE-SIGHT® oximeters, during shoulder surgery in the beach chair position.

(iii) Assess the relationships between cerebral oxygen desaturation during shoulder surgery in the BCP and variables including mean arterial pressure, incidence of nausea/vomiting, duration of hospital stay, BMI, hypertension and adverse events.

RESEARCH QUESTION There are three research questions correlating with the three research aims; (i) Is cerebral desaturation during shoulder surgery associated with POCD? (ii) Do the FORE-SIGHT® and INVOS™ 5100 devices vary in their measurement of cerebral oxygenation during shoulder surgery in the BCP? (iii) Is there a relationship between cerebral desaturation events during shoulder surgery in the BCP and variables including mean arterial blood pressure, post-operative nausea/vomiting, length of hospital stay, BMI, hypertension and any adverse events?

NULL HYPOTHESES The three null hypotheses are; (i) Cerebral desaturation as measured using cerebral oximetry is not related to POCD after shoulder surgery in the BCP.

(ii) There is no significant difference between the INVOS™ 5100 and the FORE-SIGHT® monitors assessment of cerebral oxygenation during shoulder surgery in the BCP.

(iii) There is no relationship between cerebral desaturation events during shoulder surgery in the BCP and variables including mean arterial blood pressure, the frequency of post-operative nausea/vomiting, length of hospital stay, BMI, hypertension and any adverse events.

PRIMARY HYPOTHESES The primary research hypotheses are; (i) Cerebral desaturation events during surgery in the BCP will be related to POCD.

(ii) The INVOS™ 5100 and the FORE-SIGHT® monitors will show no significant difference in their ability to measure cerebral oxygenation.

(iii) Cerebral desaturation events experienced during shoulder surgery in the BCP are related to a drop in mean arterial blood pressure, an increased likelihood of post-operative nausea and vomiting, greater length of hospital stay, a higher BMI, hypertension and greater frequency of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Receiving treatment primarily by, but not restricted to, one of the Primary investigators for a shoulder condition that requires surgery in the BCP.
* Over 18 years of age
* Able to read and speak English

Exclusion Criteria:

* Under 18 years of age
* Pregnant women
* Pre-operative Mini-Mental State Examination (MMSE) < 24
* Pre-existing cerebrovascular disease as reported by the assessing medical consultant and recorded in patient charts
* Orthostatic hypotension
* American Society of Anaesthesiologists (ASA) physical status III, IV and V*
* History of drug and/or alcohol abuse
* Neurological disease (e.g. previous stroke)
* Significant mood and anxiety disorders as determined by treating consultant.
* Any other condition, which in the opinion of the investigators, would render the patient unsuitable for participation in the study

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-05-25 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Trail making test: Delis-Kaplan Executive Function System | Baseline
  The D-KEFs Trails subtest has four trials; visual scanning, number sequencing, letter sequencing and letter number sequencing.
Trail making test: Delis-Kaplan Executive Function System | 1 day post-operative
  The D-KEFs Trails subtest has four trials; visual scanning, number sequencing, letter sequencing and letter number sequencing.
Trail making test: Delis-Kaplan Executive Function System | 8-14 days post-operative
  The D-KEFs Trails subtest has four trials; visual scanning, number sequencing, letter sequencing and letter number sequencing.
Trail making test: Delis-Kaplan Executive Function System | 6 weeks post-operative
  The D-KEFs Trails subtest has four trials; visual scanning, number sequencing, letter sequencing and letter number sequencing.
Trail making test: Delis-Kaplan Executive Function System | 3 months post-operative
  The D-KEFs Trails subtest has four trials; visual scanning, number sequencing, letter sequencing and letter number sequencing.
Single letter verbal fluency | Baseline
  This task requires the individual to spontaneously generate a list of words in 60 seconds, where the words cannot be name of places, people or other proper nouns.
Single letter verbal fluency | 1 day post-operative
  This task requires the individual to spontaneously generate a list of words in 60 seconds, where the words cannot be name of places, people or other proper nouns.
Single letter verbal fluency | 8-14 days post-operative
  This task requires the individual to spontaneously generate a list of words in 60 seconds, where the words cannot be name of places, people or other proper nouns.
Single letter verbal fluency | 6 weeks post-operative
  This task requires the individual to spontaneously generate a list of words in 60 seconds, where the words cannot be name of places, people or other proper nouns.
Single letter verbal fluency | 3 months post-operative
  This task requires the individual to spontaneously generate a list of words in 60 seconds, where the words cannot be name of places, people or other proper nouns.
Rey Auditory Verbal Learning Test | Baseline
  The RAVLT assesses immediate and delayed auditory memory recall and recognition. The task consists of 15 nouns learned over 5 trials with a free recall after each presentation. The order of presentation remaining fixed across trials (List A). At the end of the 5th trial an interference list of 15 words is presented (List B), following a free recall of that list. Immediately after this, delayed recall of the first list is tested. Following a 20-minute delay, delayed recall and recognition of the first word list is assessed.
Rey Auditory Verbal Learning Test | 1 day post-operative
  The RAVLT assesses immediate and delayed auditory memory recall and recognition. The task consists of 15 nouns learned over 5 trials with a free recall after each presentation. The order of presentation remaining fixed across trials (List A). At the end of the 5th trial an interference list of 15 words is presented (List B), following a free recall of that list. Immediately after this, delayed recall of the first list is tested. Following a 20-minute delay, delayed recall and recognition of the first word list is assessed.
Rey Auditory Verbal Learning Test | 8-14 days post-operative
  The RAVLT assesses immediate and delayed auditory memory recall and recognition. The task consists of 15 nouns learned over 5 trials with a free recall after each presentation. The order of presentation remaining fixed across trials (List A). At the end of the 5th trial an interference list of 15 words is presented (List B), following a free recall of that list. Immediately after this, delayed recall of the first list is tested. Following a 20-minute delay, delayed recall and recognition of the first word list is assessed.
Rey Auditory Verbal Learning Test | 6 weeks post-operative
  The RAVLT assesses immediate and delayed auditory memory recall and recognition. The task consists of 15 nouns learned over 5 trials with a free recall after each presentation. The order of presentation remaining fixed across trials (List A). At the end of the 5th trial an interference list of 15 words is presented (List B), following a free recall of that list. Immediately after this, delayed recall of the first list is tested. Following a 20-minute delay, delayed recall and recognition of the first word list is assessed.
Rey Auditory Verbal Learning Test | 3 months post-operative
  The RAVLT assesses immediate and delayed auditory memory recall and recognition. The task consists of 15 nouns learned over 5 trials with a free recall after each presentation. The order of presentation remaining fixed across trials (List A). At the end of the 5th trial an interference list of 15 words is presented (List B), following a free recall of that list. Immediately after this, delayed recall of the first list is tested. Following a 20-minute delay, delayed recall and recognition of the first word list is assessed.
Letter-Number Sequencing (from Wechsler Adult Intelligence Scale, 4th edition) | Baseline
  The examinee is verbally presented with a combination of numbers and letters or increasing amounts. The examinee is required to recall the numbers in ascending order then letters in alphabetical order.
Letter-Number Sequencing (from Wechsler Adult Intelligence Scale, 4th edition) | 1 day post-operative
  The examinee is verbally presented with a combination of numbers and letters or increasing amounts. The examinee is required to recall the numbers in ascending order then letters in alphabetical order.
Letter-Number Sequencing (from Wechsler Adult Intelligence Scale, 4th edition) | 8-14 days post-operative
  The examinee is verbally presented with a combination of numbers and letters or increasing amounts. The examinee is required to recall the numbers in ascending order then letters in alphabetical order.
Letter-Number Sequencing (from Wechsler Adult Intelligence Scale, 4th edition) | 6 weeks post-operative
  The examinee is verbally presented with a combination of numbers and letters or increasing amounts. The examinee is required to recall the numbers in ascending order then letters in alphabetical order.
Letter-Number Sequencing (from Wechsler Adult Intelligence Scale, 4th edition) | 3 months post-operative
  The examinee is verbally presented with a combination of numbers and letters or increasing amounts. The examinee is required to recall the numbers in ascending order then letters in alphabetical order.

SECONDARY OUTCOMES:
Cerebral desaturation events (INVOS) | Intra-operative
  Cerebral desaturation will be defined as a decrease in regional cerebral oxygen saturation greater than, or equal to 20% from baseline or a fall below 50% absolute.
Cerebral desaturation events (FORE-SIGHT) | Intra-operative
  Cerebral desaturation will be defined as a decrease in regional cerebral oxygen saturation greater than, or equal to 20% from baseline or a fall below 50% absolute.
Mean arterial pressure | Intra-operative
  Mean arterial blood pressure (mmHg)
Body Mass Index | Baseline
  Patient Body Mass Index (BMI)
Hypertension | Baseline
  Patient-reported hypertension
Nausea and vomiting within 48 hours | 1 day, 8-14 days
  Patient-reported nausea and vomiting
Duration of hospital stay | 8-14 days
  Patient duration of hospital stay
Adverse events | Intra-operative
  Any adverse events arising during the trial will be closely monitored and followed up until the resolution of symptoms. These will be checked at each assessment stage and recorded on a data collection form.
Adverse events | 1 day
  Any adverse events arising during the trial will be closely monitored and followed up until the resolution of symptoms. These will be checked at each assessment
Adverse events | 8-14 days
  Any adverse events arising during the trial will be closely monitored and followed up until the resolution of symptoms. These will be checked at each assessment
Adverse events | 6 weeks
  Any adverse events arising during the trial will be closely monitored and followed up until the resolution of symptoms. These will be checked at each assessment
Adverse events | 3 months
  Any adverse events arising during the trial will be closely monitored and followed up until the resolution of symptoms. These will be checked at each assessment

OTHER OUTCOMES:
Depression Anxiety and Stress Scale-21 | Baseline, 1 day, 8-14 days, 6 weeks, 3 months
  The DASS-21 has 21 questions that index the level of depression, anxiety and stress an individual has experienced in the preceding week.
Social Relationships and Support Scale | Baseline, 1 day, 8-14 days, 6 weeks, 3 months
  The social support measures address the issues of social process in a range different clinical populations.
Loneliness Scale | Baseline, 1 day, 8-14 days, 6 weeks, 3 months
  A standardised 3-item Loneliness scale, comprised of items from the well-validated University of California, Los Angeles (UCLA) Loneliness scale.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Ross, MBBS, Principal Investigator — Director
Locations (1):
- Brisbane Hand and Upper Limb Research Institute, Brisbane Private Hospital, Brisbane, Queensland, Australia

IPD SHARING:
Plan to Share IPD: Yes
Deidentified cerebral oximeter data acquisition files will be made available to the equipment manufacturers (Medtronic, CASMED) at the conclusion of the study.

REFERENCES:
- See also: Brisbane Hand and Upper Limb Research Institute — http://www.upperlimb.com

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2018-06-01): https://cdn.clinicaltrials.gov/large-docs/45/NCT03036345/Prot_ICF_000.pdf